CLINICAL TRIAL: NCT04341974
Title: Perioperative Use of Serum Creatinine and Postoperative Acute Kidney Injury: an Observational, Monocentric, Retrospective Study to Explore Physicians' Perception and Practice.
Brief Title: Perioperative Use of Serum Creatinine and Postoperative Acute Kidney Injury
Acronym: CreaPeriop
Status: Completed | Type: Observational
Sponsor: Careggi Hospital (Other)
Responsible Party: Principal Investigator, Gianluca Villa, MD, clinical researcher, Careggi Hospital
Other Study IDs: CEAVC 13881/2018
Record Dates: First submitted 2020-04-08; First posted 2020-04-10 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Surgery; Malignancy; Acute Kidney Injury; Cronich Kidney Disease
Keywords: serum creatinine; kidney dysfunction
MeSH Terms: conditions — Neoplasms; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- surgical patients: Adult patients undergoing major elective general abdominal surgery for ontological disease
  Interventions: Diagnostic Test: Serum creatinine

INTERVENTIONS:
Diagnostic Test: Serum creatinine — Will be described: 1) the number of patients actually screened with postoperative serum creatinine and 2) the number of patients actually screened with the same parameter at the long-term after surgery

SUMMARY:
The perioperative approach adopted in a cohort of adult oncological patients undergoing major abdominal surgery will be described. In particular, the physician's attitude toward use of sCr for identification of patients at risk for PO-AKI will be described, as well as the patients who should be reassessed in the long term for progression toward CKD. The incidence and risk factors associated with PO-AKI and renal function deterioration within a year postoperatively will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Scheduled for elective surgery
* Surgery for oncological disease

Exclusion Criteria:

* Patients undergoing postoperative chemotherapy
* Patients who died within 12 month after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients were older than 18 years, underwent surgery under general anesthesia for oncological disease who underwent major elective general abdominal surgery from November 2016 to February 2017 at the Department of Anaesthesia of Careggi Hospital
Sampling Method: Non-Probability Sample
Enrollment: 423 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Adoption of serum creatinine as marker of acute kidney injury postoperively | 3rd postoperative day
  Number of actual patients screened postoperatively

SECONDARY OUTCOMES:
Incidence of acute kidney injury | 3rd postoperative day
  Number of patients with a postoperative diagnostic increase of serum creatinine, in accordance with KDIGO guidelines
Adoption of serum creatinine as marker of long term kidney dysfunction | 12 month after surgery
  Number of actual patients screened at the long term
Incidence of long term kidney dysfunction | 12 month after surgery
  Number of patients with a long term reduction in GFR greater than 10 ml/min with respect to the baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria Careggi, Florence, Italy

IPD SHARING:
Plan to Share IPD: No
IPD will be not shared

REFERENCES:
- [Derived] Villa G, De Rosa S, Scire Calabrisotto C, Nerini A, Saitta T, Degl'Innocenti D, Paparella L, Bocciero V, Allinovi M, De Gaudio AR, Ostermann M, Romagnoli S. Perioperative use of serum creatinine and postoperative acute kidney injury: a single-centre, observational retrospective study to explore physicians' perception and practice. Perioper Med (Lond). 2021 May 25;10(1):13. doi: 10.1186/s13741-021-00184-6. PMID 34030728